CLINICAL TRIAL: NCT00821418
Title: Assessment of the Safety and the Effect on Patients With COPD of Treatment With PulseHaler™ - a Novel Device for Pulsating Positive Expiratory Pressure Ventilation
Brief Title: Assessment of Treatment With PulseHaler on Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Respinova LTD (Industry)
Responsible Party: Yuval Avni, Respinova
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PLS-01
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- PulsHaler first (Experimental)
  Interventions: Device: PulseHaler treatment
- Placebo first (Placebo Comparator)
  Interventions: Device: CPAP treatment (through a deactivated version of PulsHaler)

INTERVENTIONS:
Device: PulseHaler treatment — treatment is for two weeks, 3 times per day
  Arms: PulsHaler first
Device: CPAP treatment (through a deactivated version of PulsHaler) — treatment is for two weeks, 3 times per day
  Arms: Placebo first

SUMMARY:
The purpose of the study is to assess the safety and the effect of treatment by PulseHaler™ on patients with COPD, as measured by the change from baseline in full pulmonary functions, oxygen saturation, exercise tolerance and health related quality of life; and to assess the ease of use of PulseHaler™ by the patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Diagnosis established for at least 1 year;
* Post-bronchodilator FEV1/FVC < 0.7
* Post bronchodilator FEV1 <70% predicted
* Age: 40 years or older
* Smoking cigarettes, at least 10PY
* Patient signed the informed consent form

Exclusion Criteria:

* Bullous Emphysema (ruled out by recent CT)
* Hospitalization due to exacerbation of COPD within the last 3 months
* Upper respiratory infection and/or exacerbation of COPD in the last 4 weeks
* Systemic steroid treatment in the last 4 weeks
* Women at the age of fertility, who are pregnant, or plan pregnancy, or do not use contraceptive.
* Severe cardiac disease, e.g., CHF grade 3 or higher
* Acute MI within last 3 months
* CABG within last 3 months
* Other severe systemic disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Pulmonary function tests | Within 2 hours from first treatment, and after 2 weeks of treatment
Six minute walk test | Within 2 hours from first treatment, and after 2 weeks of treatment
Health related quality of life | Within 2 hours from first treatment, and after 2 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Fridlender ZG, Arish N, Laxer U, Berkman N, Leibovitz A, Fink G, Breuer R. Randomized controlled crossover trial of a new oscillatory device as add-on therapy for COPD. COPD. 2012 Dec;9(6):603-10. doi: 10.3109/15412555.2012.748625. Epub 2012 Dec 6. PMID 23215916